CLINICAL TRIAL: NCT06828172
Title: Local or Systemic Vascular Effects: Mechanisms Related to Arm Crank Exercise - Comparison Between Individuals With and Without PAD
Brief Title: Local or Systemic Effects: Mechanisms Related to Arm Crank Exercise - Comparison Between Individuals With and Without PAD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Collaborators: University of Sao Paulo (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Marilia de Almeida Correia, PhD, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EB_PADvsHealth
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Peripheral Arterial Disease
Keywords: Intermittent claudication; Exercise; Vascular function
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm crank exercise (Experimental): In the arm-cranking condition, the patients will perform fifteen bouts of two minutes of arm-cranking with an interval of two minutes between bouts, at an intensity equivalent to 13-15 on Borg's subjective perceived exertion scale. The condition will have a total of sixty minutes of duration.
  Interventions: Behavioral: Exercise
- Control Condition (Sham Comparator): The control condition will consist of resting in the standing position for thirty minutes. The patients will be instructed to rest in the sitting position for two minutes at periods equivalent to the intervals from the exercise conditions, totalling sixty minutes of duration.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Two conditions will be tested: Arm-cranking and control condition.

SUMMARY:
INTRODUCTION: Exercise with an arm ergometer (EB) overcomes the main barrier to physical exercise in patients with Peripheral Artery Disease (PAD), leg pain during walking. Due to its aerobic nature, this type of exercise can cause systemic changes in the regulatory mechanisms of vasodilation. In other words, it provides vascular benefits in the most affected arterial beds in the PAD population. OBJECTIVE: To analyze local and systemic vascular responses, as well as cell signaling pathways after an EB exercise session in patients with PAD and their peers without PAD. METHODS: 24 patients with PAD and 24 individuals without PAD will be recruited, matched by sex and age. Participants will undergo two experimental sessions in approved order (EB and control). The EB session will consist of 15 cycles of 2 min of exercise with an intensity equivalent to 13-15 on the Borg scale of perceived exertion. Before and after the experimental sessions, the vascular function of the brachial and femoral arteries, blood indicators of vasodilation and calf muscle oxygenation will be evaluated. To analyze the acute effect between groups on cardiovascular parameters, a three-way analysis of variance will be performed, taking as factors disease (presence vs. absence), session (EB vs. Control) and time (pre vs. post). In all analyses, when a significant effect is selected, the Bonferroni or Newman-Keuls post-hoc test will be used. For all analyses, a value of P<0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* If female, must be postmenopausal without hormone replacement therapy;
* Non-smokers;
* With a body mass index (BMI) not exceeding 30 kg/m²;
* With calf skinfold thickness below 20 mm, due to the interference of adiposity in the penetration of light from the NIRS probe, and oxygen saturation in the finger >95% to ensure that impaired pulmonary gas exchange does not affect oxygen saturation measurements in the calf;
* Not using classic antioxidants or vitamin supplements; and
* Physically capable of performing an exercise session.
* For the group of participants with PAD, in addition to the criteria mentioned above, they must have a confirmed diagnosis of the disease, characterized by an ankle-brachial index (ABI) lower than 0.90 in one or both legs, exhibit symptoms of claudication during walking, and be physically capable of performing an exercise session to participate in the project.

Exclusion Criteria:

* Only participants who discontinue their participation in the study protocol will be excluded from the sample

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Calf Muscle Oxygen Saturation (%) | Just before, during 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30 minutes of exercise, and after 10 minutes of exercise.
  The parameters of calf muscle oxygenation will be collected using the non-invasive Near-Infrared Spectroscopy (NIRS) technique, with an NIRS spectrometer and a dedicated laptop computer. The NIRS sensor will be placed on the calf region, on the leg with the lower ankle brachial index, at the level of the largest calf circumference. The equipment will be programmed for continuous recording throughout the experimental session, covering the pre-exercise, during exercise with arm ergometer, and post-exercise periods.

SECONDARY OUTCOMES:
Change from baseline in vascular function post-exercise in the brachial and femoral arteries (%). | Before and after 40 minutes of exercise.
  Vascular function will be measured in the supine position by the flow-mediated dilation (FMD) technique, through Doppler ultrasonography.
Oxyhemoglobin (micromol) | Just before, during 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30 minutes of exercise, and after 10 minutes of exercise.
  The parameters of calf muscle oxygenation will be collected using the non-invasive Near-Infrared Spectroscopy (NIRS) technique, with an NIRS spectrometer and a dedicated laptop computer. The NIRS sensor will be placed on the calf region, on the leg with the lower ankle brachial index, at the level of the largest calf circumference. The equipment will be programmed for continuous recording throughout the experimental session, covering the pre-exercise, during exercise with arm ergometer, and post-exercise periods.
Deoxyhemoglobin (micromol) | Just before, during 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30 minutes of exercise, and after 10 minutes of exercise.
  The parameters of calf muscle oxygenation will be collected using the non-invasive Near-Infrared Spectroscopy (NIRS) technique, with an NIRS spectrometer and a dedicated laptop computer. The NIRS sensor will be placed on the calf region, on the leg with the lower ankle brachial index, at the level of the largest calf circumference. The equipment will be programmed for continuous recording throughout the experimental session, covering the pre-exercise, during exercise with arm ergometer, and post-exercise periods.
Total hemoglobin (micromol) | Just before, during 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30 minutes of exercise, and after 10 minutes of exercise.
  The parameters of calf muscle oxygenation will be collected using the non-invasive Near-Infrared Spectroscopy (NIRS) technique, with an NIRS spectrometer and a dedicated laptop computer. The NIRS sensor will be placed on the calf region, on the leg with the lower ankle brachial index, at the level of the largest calf circumference. The equipment will be programmed for continuous recording throughout the experimental session, covering the pre-exercise, during exercise with arm ergometer, and post-exercise periods.
Nitric oxide production markers (micromol) | Before and after 5 minutes of exercise.
  Before and after the sessions, a venous blood sample (10 mL) will be collected in tubes containing Ethylenediaminetetraacetic Acid (EDTA). Plasma will be immediately obtained after refrigerated centrifugation and used for the determination of thiobarbituric acid reactive substances (TBARS), nitrite, and nitrate (Griess test, Sigma Aldrich), as well as for biochemical analyses of lipids (cholesterol, triglycerides, High-Density Lipoprotein (HDL) cholesterol, and Low-Density Lipoprotein (LDL) cholesterol calculation) and glucose levels. Glycated hemoglobin will be determined in whole blood by high-performance liquid chromatography. Cultured human umbilical vein endothelial cells (HUVEC) will be incubated with 0.2% plasma obtained from all individuals for different time intervals. Indicators of nitric oxide production will be determined in the cells (cGMP concentration and endothelial nitric oxide synthase [eNOS] expression) and in the culture medium (nitrite/nitrate concentration).

CONTACTS AND LOCATIONS:
Overall Officials: Marilia A Correia, PhD, Principal Investigator — University of Nove de Julho
Locations (1):
- University Nove de Julho, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Individual data may be disclosed upon contact with the principal investigator.
Supporting Information: Study Protocol, SAP, CSR